CLINICAL TRIAL: NCT01308476
Title: Assessment if a Daily SMS (Short Message System) Reminder Improves the Adherence of COPD Patients to Therapy With Spiriva® 18 Microgram
Brief Title: SMS Reminder to Assess Adherence
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.474
Record Dates: First submitted 2011-03-01; First posted 2011-03-04 (Estimated); Results first posted 2012-12-21 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Control Groups

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- SMS group
  Interventions: Procedure: SMS reminder
- control group
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: SMS reminder — daily SMS in the SMS group to remind of treatment with tiotropium
  Groups: SMS group
Procedure: control group — no daily SMS to remind of treatment with tiotropium
  Groups: control group

SUMMARY:
6 months open label non-interventional observational study acc to § 4, section 23 and § 67, section 6 German Medicines Act with two parallel groups

1. the SMS group receiving a daily SMS - a reminder to inhale Spiriva® 18 Microgram
2. the control group not receiving a daily SMS reminder

DETAILED DESCRIPTION:
Purpose:

Study Design:

observational

ELIGIBILITY:
Inclusion criteria:

* Chronic obstructive pulmonary disease (COPD) patients requiring long-acting bronchodilators according to approved Summary of Product Characteristics (SPC) and guidelines
* User of mobile phone

Exclusion criteria:

- Patients presenting with the general and specific contraindications listed in the Patient Information Leaflet and the SPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- Germany (5):
  - Boehringer Ingelheim Investigational Site 1, Berlin
  - Boehringer Ingelheim Investigational Site 2, Cottbus
  - Boehringer Ingelheim Investigational Site 3, Hamburg
  - Boehringer Ingelheim Investigational Site 4, Koblenz
  - Boehringer Ingelheim Investigational Site 5, Lübeck

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who participated in this study had to have access to a mobile phone since a SMS (short message service) / IVR (interactive voice response) system was used to remind to medication intake and to evaluate the adherence to Spiriva HandiHaler.
Pre-assignment Details: Non-interventional controlled pilot study with two parallel groups.
Groups:
- SMS Reminder Group: Patients receive a daily SMS to remind them to inhale Spiriva 18 mcg by using HandiHaler.
- Control Group: Control group with same medication but not receiving reminder SMS.
Period: Overall Study
Arm/Group | SMS Reminder Group | Control Group
Started | 48 (Entered and treated.) | 47 (Entered and treated.)
Completed | 45 | 45
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMS Reminder Group | Control Group | Total
Number analyzed (Participants) | 48 | 47 | 95
Age Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (7.3) | 63.2 (8.1) | 62.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 33 | 30 | 63

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Spiriva HandiHaler Over Time
Description: Adherence was defined as percentage of documented applications of Spiriva HandiHaler as compared to the regularly planned seven applications during the week before questioning the patients. Patients in the SMS reminder group and in the control group were asked via SMS how often they had used Spiriva HandiHaler during the last week and were requested to call the IVR system to provide their response. Baseline was defined as week 4.
Time Frame: Baseline, Week 8, Week 12, Week 16, Week 20 and Week 24
Population: Full Analysis Set (FAS) is defined as all treated patients who additionally met the study diagnosis (Chronic Obstructive Pulmonary Disease (COPD) requiring long-acting anticholinergics) and who had evaluable data in at least one effectiveness endpoint.
  Only subjects who responded to the SMS/ IVR system were considered in this analysis.
Measure: Mean (Standard Deviation); unit: Percentage of applications
Arm/Group | SMS Reminder Group | Control Group
Number analyzed (Participants) | 28 | 26
Percentage of applications
  Baseline | 99.0 (5.4) | 96.2 (12.5)
  Week 8 (N=28, 29) | 99.5 (2.7) | 99.5 (2.7)
  Week 12 (N=20, 30) | 100.0 (0.0) | 98.6 (7.8)
  Week 16 (N=25, 29) | 100.0 (0.0) | 96.1 (14.2)
  Week 20 (N=27, 29) | 100.0 (0.0) | 95.1 (18.8)
  Week 24 (N=26, 30) | 99.5 (2.8) | 95.7 (18.4)

2. Secondary Outcome: Change From Baseline in Adherence to Spiriva HandiHaler Over Time
Description: as for outcome 1
Time Frame: Week 8, Week 12, Week 16, Week 20 and Week 24
Population: FAS. Only subjects who responded to the SMS/ IVR system were considered in this analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | SMS Reminder Group | Control Group
Number analyzed (Participants) | 23 | 23
Percent change
  Week 8 | 0.6 (3.0) | 3.7 (12.3)
  Week 12 (N=15, 23) | 0.0 (0.0) | 2.5 (16.5)
  Week 16 (N=20, 20) | 0.0 (0.0) | 0.7 (22.0)
  Week 20 (N=20, 21) | 0.0 (0.0) | -1.4 (11.0)
  Week 24 (N=21, 23) | 0.0 (0.0) | -1.2 (9.5)

3. Secondary Outcome: Response Rate Regarding Adherence
Description: Adherence was dichotomised into yes and no at the end of study depending on whether the percentage of adherence was at least 80 percent or less than 80 percent, respectively. Patients who did not respond to the SMS/ IVR system to provide information about the actual number of inhalations were considered with 0 percent adherence.
Time Frame: 24 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | SMS Reminder Group | Control Group
Number analyzed (Participants) | 47 | 45
Percentage of participants
  yes (adherent) | 55.3 | 64.4
  no (not adherent) | 44.7 | 35.6

4. Secondary Outcome: Patients Compliance With SMS System
Description: Compliance was defined as the percentage of patients answers to the IVR system as compared to the number of SMS automatically sent to the patients by the SMS/ IVR system asking for the number of Spiriva HandiHaler applications.
Time Frame: 24 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Percentage of participants answers
Arm/Group | SMS Reminder Group | Control Group
Number analyzed (Participants) | 47 | 45
Percentage of participants answers | 55.0 (39.8) | 64.1 (38.3)

5. Secondary Outcome: Patients Assessment of Usefulness of the SMS System
Description: Only patients in the SMS reminder group were asked to assess the usefulness of the SMS system by the categories very helpful, helpful and not helpful.
Time Frame: Visit 2 (12 weeks) and visit 3 (24 weeks)
Population: FAS for SMS reminder group only
Measure: Number; unit: Percentage of participants
Arm/Group | SMS Reminder Group | Control Group
Number analyzed (Participants) | 47 | 0
Percentage of participants
  Very helpful (week 12) | 12.8 |
  Helpful (week 12) | 61.7 |
  Not helpful (week 12) | 23.4 |
  Missing (week 12) | 2.1 |
  Very helpful (week 24), N=45 | 8.9 |
  Helpful (week 24), N=45 | 53.3 |
  Not helpful (week 24), N=45 | 33.3 |
  Missing (week 24), N=45 | 4.4 |

6. Secondary Outcome: Physicians Assessment of Usefulness of the SMS System
Description: Only physicians of patients in the SMS reminder group were asked to assess the usefulness of the SMS system by the categories very helpful, helpful and not helpful.
Time Frame: Visit 2 (12 weeks) and visit 3 (24 weeks)
Population: FAS for SMS reminder group only
Measure: Number; unit: Percentage of participants
Arm/Group | SMS Reminder Group | Control Group
Number analyzed (Participants) | 47 | 0
Percentage of participants
  Very helpful (week 12) | 6.4 |
  Helpful (week 12) | 87.2 |
  Not helpful (week 12) | 6.4 |
  Missing (week 12) | 0.0 |
  Very helpful (week 24), N=45 | 11.1 |
  Helpful (week 24), N=45 | 80.0 |
  Not helpful (week 24), N=45 | 6.7 |
  Missing (week 24), N=45 | 2.2 |

7. Secondary Outcome: Physicians Recommendation of the SMS System
Description: Only physicians of patients in the SMS reminder group were asked if they would recommend the SMS system (no, yes, don't know)
Time Frame: Visit 2 (12 weeks) and visit 3 (24 weeks)
Population: FAS for SMS reminder group only
Measure: Number; unit: Percentage of participants
Arm/Group | SMS Reminder Group | Control Group
Number analyzed (Participants) | 47 | 0
Percentage of participants
  No (week 12) | 8.5 |
  Yes (week 12) | 70.2 |
  Don't know (week 12) | 21.3 |
  No (week 24), N=45 | 8.9 |
  Yes (week 24), N=45 | 64.4 |
  Don't know (week 24), N=45 | 26.7 |

8. Secondary Outcome: Patients Satisfaction With SMS System
Description: Only patients in the SMS group were asked to assess their satisfaction with the SMS system by assigning German school grades 1=very good, 2=good, 3=satisfactory, 4=sufficient, 5=deficient, 6=insufficient.
Time Frame: Visit 2 (12 weeks) and visit 3 (24 weeks)
Population: FAS for SMS reminder group only
Measure: Number; unit: Percantage of participants
Arm/Group | SMS Reminder Group | Control Group
Number analyzed (Participants) | 47 | 0
Percantage of participants
  Very good (week 12) | 23.4 |
  Good (week 12) | 42.6 |
  Satisfactory (week 12) | 21.3 |
  Sufficient (week 12) | 6.4 |
  Deficient (week 12) | 2.1 |
  Insufficient (week 12) | 4.3 |
  Very good (week 24), N=45 | 15.6 |
  Good (week 24), N=45 | 37.8 |
  Satisfactory (week 24), N=45 | 28.9 |
  Sufficient (week 24), N=45 | 11.1 |
  Deficient (week 24), N=45 | 4.4 |
  Insufficient (week 24), N=45 | 2.2 |

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | SMS Reminder Group | Control Group
Serious Adverse Events (participants affected / at risk) | 2/48 | 2/47
Other Adverse Events (participants affected / at risk) | 0/48 | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SMS Reminder Group (N=48) | Control Group (N=47)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.